CLINICAL TRIAL: NCT00597610
Title: Evaluating The Response to Pre-Operative Chemotherapy and/or Radiation Therapy For Rectal Cancer Using Three-Dimension Transrectal Ultrasound (3-D TRUS) - A Pilot Project
Brief Title: Evaluating The Response to Pre-Operative Chemotherapy and/or Radiation Therapy For Rectal Cancer Using Three-Dimension Transrectal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-127
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Rectal Cancer
Keywords: Rectum; Rectal
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Transrectal ultrasound 3-D (TRUS)

INTERVENTIONS:
Other: Transrectal ultrasound 3-D (TRUS) — Transrectal ultrasound (TRUS) is widely accepted as an accurate and effective technique for staging of rectal cancer. The decision to administer pre-operative chemotherapy/radiation therapy is often made based on the results of the TRUS. Three-dimensional TRUS (3-D TRUS) is a new modality that provides all of the information of traditional TRUS as well as the ability to provide three dimensional views of the tumor.

SUMMARY:
Traditional transrectal ultrasound (TRUS) is a technique used to help determine the stage of rectal cancer. All patients at Memorial Sloan-Kettering Cancer Center with rectal cancer have an ultrasound at the beginning of their treatment to accurately determine the depth of penetration (how deep into the rectal wall the tumor goes) and lymph node involvement of their tumor. This information helps determine the best way to treat the patient's disease. Three-dimensional TRUS (3-D TRUS) is a new form of ultrasound that gives us all of the information of traditional ultrasound in addition to being able to view the tumor in 3-dimensions. This image can be stored and analyzed to evaluate the tumor size and volume as well as determine the unique shape of the tumor. Chemoradiotherapy before surgery is considered standard of care for most rectal cancers.

Currently, there is no accurate way to determine whether or not the tumor has responded to the pre-operative radiation therapy. The purpose of this study is to evaluate the response of rectal cancer to pre-operative chemotherapy and/or radiation therapy using 3-D TRUS to measure the volume of the tumor before and after chemoradiotherapy.

DETAILED DESCRIPTION:
Transrectal ultrasound (TRUS) is widely accepted as an accurate and effective technique for staging of rectal cancer. The decision to administer pre-operative chemotherapy/radiation therapy is often made based on the results of the TRUS. The greatest limitation of TRUS is its operator-dependence. Three-dimensional TRUS (3-D TRUS) is a new modality that provides all of the information of traditional TRUS as well as the ability to provide three dimensional views of the tumor. This provides greater detail regarding the configuration of the tumor as well as the ability to calculate tumor volume. The results of 3-D TRUS are interpreted after the study and thus, operator-dependence is reduced. There are no currently accepted techniques that allow for objective and accurate assessment of a rectal tumor's response to pre-operative treatment short of post-operative pathologic evaluation. Our objectives are to evaluate the ability of 3-D TRUS to quantify the tumor's response to pre-operative radiation therapy and/or chemotherapy and to correlate these findings with post-operative pathologic examination of the specimen. These objectives can be accomplished with 2 ultrasounds, one before treatment and one before surgery. All patients with biopsy-proven (with pathology confirmed at MSKCC) rectal cancer are eligible for the study. The size, volume and depth of penetration and lymph node involvement will all be assessed during both ultrasound examinations. Our findings will then be compared to those found at post-operative pathologic examination. These data will then be analyzed to determine if 3-D TRUS was accurate in predicting the tumor's response to preoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven rectal cancer (path confirmed at MSKCC)
* able to provide consent for 3-D TRUS
* eligible for pre-operative chemotherapy and/or radiation therapy

Exclusion Criteria:

* unable to provide informed consent
* unable to tolerate 3-D TRUS either pre- or post-chemo/RT
* unable to tolerate full course of chemotherapy and/or radiation therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To measure the response of primary rectal cancer to neoadjuvant chemotherapy and/or radiation therapy using 3-D TRUS | 6 years

SECONDARY OUTCOMES:
To correlate these findings with post-operative pathologic examination | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weiser, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org